CLINICAL TRIAL: NCT05356286
Title: Recording of Intraoperative Spinal Cord Stimulation and Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Professor, Neurosurgery, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-000043
Record Dates: First submitted 2022-04-22; First posted 2022-05-02 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cervical Stenosis; Disk, Herniated; Spondylosis
MeSH Terms: conditions — Intervertebral Disc Displacement; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Electrical Stimulation group (Experimental): Epidural Electrical Stimulation of the Cervical Spinal Cord
  Interventions: Device: epidural electrical stimulation

INTERVENTIONS:
Device: epidural electrical stimulation — Electrical spinal cord stimulation will be used to modulate respiratory function during general anesthesia.

SUMMARY:
Opioid overdose suppresses brainstem respiratory circuits, causes apnea, and may result in death. Epidural electrical stimulation (EES) at the cervical spinal cord facilitated motor activity in rodents and humans, and we hypothesized that EES of the cervical spinal cord could antagonize opioid-induced respiratory depression in humans. In this study, we will stimulate the spinal cord during surgery and assess its effects on respiratory function in human patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patients undergoing brain or spinal cord surgery where spinal neuromonitoring is utilized.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-01-21 (Actual); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Change in respiratory frequency | During intraoperative surgery during stimulation and within 2 minutes after stimulation
  Increase or decrease in respiratory frequency of 20% during or after stimulation
Change in respiratory tidal volume | During intraoperative surgery during stimulation and within 2 minutes after stimulation
  Increase or decrease in respiratory tidal volume of 20% during or after stimulation

SECONDARY OUTCOMES:
Change in heart rate | During intraoperative surgery during stimulation and within 2 minutes after stimulation
  Increase or decrease in heart rate of 20% during or after stimulation
Change in blood pressure | During intraoperative surgery during stimulation and within 2 minutes after stimulation
  Increase or decrease in blood pressure of 20% during or after stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No